CLINICAL TRIAL: NCT07191184
Title: Identification of Obstacles and Levers to the Outpatient Care of Patients in Terminal Palliative Situations: Exploratory Study Among General Practitioners in Bas-Rhin
Brief Title: Identification of Obstacles and Levers to the Outpatient Care of Patients in Terminal Palliative Situations
Acronym: PTPS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9303
Record Dates: First submitted 2025-03-27; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: End of Life
Keywords: Palliative care; Terminal palliative situations
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
80% of patients wish to die at home. The number of deaths will increase in the coming years due to the aging population. The general practitioner (GP) is at the center of this care. Despite national plans for the development of palliative care, dying at home remains complicated. The difficulties described and known are organizational (workload) and linked to the doctor's experience with the suffering of the patient and their family. Many studies have been conducted in hospital settings, and the solutions developed are often not very accessible to GP. Conducting a study on this subject will allow us to take stock of this outpatient care provided by general practitioners following numerous changes that have occurred in recent years, both in terms of palliative care teaching and in terms of modifications to the care offered.

ELIGIBILITY:
Inclusion Criteria:

* General physician based in Bas-Rhin
* Agreeing to participate in the research

Exclusion Criteria:

* Refusing to participate in the research
* Replacement physician, specialist physician, based outside Bas-Rhin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General physician based in Bas-Rhin agreeing to participate in the research
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Identify barriers to outpatient care for terminally ill palliative patients by general practitioners in the Bas Rhin region. | At 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de soins Palliatifs - CHU de Strasbourg - France, Strasbourg, France